CLINICAL TRIAL: NCT05493254
Title: Hybrid Type 1 Effectiveness-Implementation Trial of a Proactive Smoking Cessation Electronic Visit for Scalable Delivery Via Primary Care
Brief Title: Enhancing Smoking Cessation Via Telehealth Options in Primary Care
Acronym: E-STOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Dahne, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00113308; R01CA258669 (NIH)
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking cessation electronic visit (e-visit) (Experimental): This group will be sent 1) an invitation to complete an electronic visit (e-visit) focused on cigarette smoking and 2) an invitation to complete a follow-up e-visit one-month after the initial e-visit.
  Interventions: Behavioral: Smoking cessation e-visit
- Treatment as usual (TAU) (Active Comparator): This group will be provided information about the state quitline and about the importance of quitting smoking and it will be recommended that they contact their PCP to schedule a medical visit to discuss quitting smoking.
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Smoking cessation e-visit — electronic visits (e-visits) for smoking cessation
  Arms: Smoking cessation electronic visit (e-visit)
Behavioral: Treatment As Usual — Information about the state quitline and about the importance of quitting smoking and a recommendation to contact one's PCP to schedule a medical visit to discuss quitting smoking.
  Arms: Treatment as usual (TAU)

SUMMARY:
The purpose of this research study is to evaluate an electronic visit (e-visit) for smoking cessation. Participants will be randomly assigned to receive either the smoking cessation e-visit or not. The e-visit will look similar to an online questionnaire asking about smoking history, motivation to quit, and preferences for medications for quitting smoking. Participants may receive a prescription for a smoking cessation medication as an outcome of the e-visit, if randomized to the e-visit group, but there is no requirement to take any medication. This study consists of questionnaires and breath samples provided at 4 separate time points throughout the study. Participation in this study will take about 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. current smoking, defined as 1+ cigarettes/day, for 20+ days out of the last 30 for the last 6+ months
2. age 18+
3. enrolled in MyChart or willing to enroll
4. possess a valid e-mail address that is checked daily
5. owner of an iOS or Android smartphone to provide remote CO
6. have a valid mailing address
7. English fluency

Exclusion Criteria:

1) Use of an FDA-approved cessation medication in the last 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who utilized smoking cessation treatment | Month 1
  Number of participants who utilized smoking cessation treatment since last assessment.
Number of participants who utilized smoking cessation treatment | Month 3
  Number of participants who utilized smoking cessation treatment since last assessment.
Number of participants who utilized smoking cessation treatment | Month 6
  Number of participants who utilized smoking cessation treatment since last assessment.
Cigarettes smoking | Month 1
  Cigarettes per day reduction greater than 50%
Cigarettes smoking | Month 3
  Cigarettes per day reduction greater than 50%
Cigarettes smoking | Month 6
  Cigarettes per day reduction greater than 50%
Quit attempts | Month 1
  Quit attempts since last contact
Quit attempts | Month 3
  Quit attempts since last contact
Quit attempts | Month 6
  Quit attempts since last contact
Seven-day point prevalence abstinence | Month 1
  Participant has not had a cigarette in the past 7 days
Seven-day point prevalence abstinence | Month 3
  Participant has not had a cigarette in the past 7 days
Seven-day point prevalence abstinence | Month 6
  Participant has not had a cigarette in the past 7 days
E-visit Acceptability | Month 1
  The e-visit will be considered acceptable if the average score on the Acceptability of Intervention Measure (AIM) is greater than or equal to 4.
E-visit Acceptability | Month 3
  The e-visit will be considered acceptable if the average score on the Acceptability of Intervention Measure (AIM) is greater than or equal to 4.
E-visit Acceptability | Month 6
  The e-visit will be considered acceptable if the average score on the Acceptability of Intervention Measure (AIM) is greater than or equal to 4.
E-visit Adoption | Month 1
  Patients prescribed a medication who obtain their medication
E-visit Adoption | Month 3
  Patients prescribed a medication who obtain their medication
E-visit Adoption | Month 6
  Patients prescribed a medication who obtain their medication

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fahey MC, Wahlquist AE, Diaz VA, Player MS, Natale N, Sterba KR, Chen BK, Hermes EDA, Carpenter MJ, Dahne J. Rationale, design, and protocol for a hybrid type 1 effectiveness-implementation trial of a proactive smoking cessation electronic visit for scalable delivery via primary care: the E-STOP trial. BMC Prim Care. 2023 Nov 29;24(1):254. doi: 10.1186/s12875-023-02205-3. PMID 38030991

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT05493254/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT05493254/ICF_001.pdf